CLINICAL TRIAL: NCT00242606
Title: Lamotrigine Versus Levetiracetam in the Initial Monotherapy of Epilepsy: An Open, Prospective, Multicenter, Randomized Phase III Study
Brief Title: Lamotrigine Versus Levetiracetam in the Initial Monotherapy of Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: UCB Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Felix Rosenow, Prof. Dr. med; PI, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LaLiMo
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Epilepsy
Keywords: Newly diagnosed epilepsy; Initial monotherapy; Levetiracetam; Lamotrigine
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine; Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Levetiracetam 2000mg/day
  Interventions: Drug: Levetiracetam
- 2 (Active Comparator): Lamotrigine
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — titrate to 200mg over 10 weeks and maintained until end of week 26
  Arms: 2
Drug: Levetiracetam — titrate to 2000mg/day over 22 days, maintain until the end of week 26
  Arms: 1

SUMMARY:
The purpose of this study is to compare the efficacy, safety and tolerance of the drugs Lamotrigine and Levetiracetam in the initial monotherapy of patients with newly diagnosed epilepsy.

DETAILED DESCRIPTION:
Epilepsy is the second most frequent neurologic disease (prevalence 0.5 % - 1 % [Brodie et al. 1997]). About 30 % of epilepsy patients (including many children) suffer from intractable seizures [Kwan & Brodie 2000]. Therefore new drugs and an expansion of permission for drugs with limited approval, respectively, are needed.

Levetiracetam is a new potent antiepileptic drug with nearly ideal pharmacokinetic properties and few side effects [Patsalos 2000], but it is approved in Germany only for add-on therapy for patients > 15 years of age with focal epilepsy.

Due to its few cognitive side effects and its efficacy, Lamotrigine is becoming standard therapy for focal and generalized epilepsy for patients from >11 years of age. Its disadvantage is the possibility of severe allergic reactions which limits the speed of dose increment.

Comparisons: Patients with newly diagnosed epilepsy are treated with either Lamotrigine or Levetiracetam. Rate of seizure-free patients in the first 6 weeks of the trial (main outcome criterion) as well as rate of seizure-free patients during the last 16 weeks and the total 26 weeks of the observation period, time until the first seizure appears, time patients take the study medication, safety and quality of life during treatment are compared.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years
* Body weight ≥ 30kg (patients 12-15 years of age) and ≥ 40kg (patients over 16 years of age), respectively
* Either one epileptic seizure with high risk of relapse (partial seizure semiology, MRI lesion or pathological focal EEG findings) or a newly diagnosed epilepsy (≥ 2 unprovoked seizures) with at least 1 seizure within the past 3 months before begin of trial participance
* Treatment with no or a maximum of one anticonvulsant drug at the time of inclusion
* Fertile women of ≥ 16 years of age must use at least one of the following contraceptives for at least one month prior to initiation of trial participance: Oral contraceptive, contraceptive diaphragm, intrauterine contraceptive device (coil), tube ligation. For girls between 12 and 15 years of age a written confirmation of sexual abstinence, given by a person having the care and custody of the child, is sufficient.
* Informed consent by the proband in written form after being informed about character, relevance and consequences of the clinical trial, and additional informed consent given by a person having the care and custody of the child for patients between 12 and 17 years of age, respectively.

Exclusion Criteria:

* Patients with non-epileptic seizures or acute symptomatic seizures whose cause can be corrected
* Patients who suffer from absence seizures or simple partial seizures without motor signs (aura) only
* Patients who had a chronic focal epilepsy or an epileptic state in their medical history
* Patients with progressive neurological, degenerative or malignant diseases which are clinically relevant from the investigator's point of view (e.g. cardiovascular or endocrinic diseases)
* Patients who have been treated with Levetiracetam or Lamotrigine before
* Patients with known manifest renal insufficiency (creatinine clearance < 80 mL/min)
* Patients with known hypersensitivity to Levetiracetam, Lamotrigine or another component of the trial drugs
* Patients who are attended by a legal guardian
* Patients suffering from a psychiatric disease or affective disorders (within the past 6 months), which had to be treated with electric convulsive therapy, tranquilizing agents, monoamine oxidase inhibitors or CNS-active sympathomimetics (e.g. methylphenidate)
* Patients who were suffering from alcohol- or drug-addiction within the past 12 months
* Pregnant or breast-feeding women
* Patients who participated in another clinical trial within the past 30 days

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2005-03; Primary Completion 2008-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Rate of seizure-free patients | in the first 6 weeks of the trial

SECONDARY OUTCOMES:
Rate of seizure-free patients | during the last 16 weeks
rate of seizure-free patients | during the total 26 weeks of the observation period
time until the first seizure appears | untin week 26
time patients take the study medication | until week 26
safety | until end of week 26
quality of life during treatment | until week 26

CONTACTS AND LOCATIONS:
Overall Officials: Felix Rosenow, M.D., Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps University Marburg Medical Center, Department of Neurology, Marburg, Germany

REFERENCES:
- [Background] Brodie MJ, Shorvon SD, Canger R, Halasz P, Johannessen S, Thompson P, Wieser HG, Wolf P. Commission on European Affairs: appropriate standards of epilepsy care across Europe.ILEA. Epilepsia. 1997 Nov;38(11):1245-50. doi: 10.1111/j.1528-1157.1997.tb01224.x. No abstract available. PMID 9579928
- [Background] Patsalos PN. Pharmacokinetic profile of levetiracetam: toward ideal characteristics. Pharmacol Ther. 2000 Feb;85(2):77-85. doi: 10.1016/s0163-7258(99)00052-2. PMID 10722121
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Derived] Rosenow F, Schade-Brittinger C, Burchardi N, Bauer S, Klein KM, Weber Y, Lerche H, Evers S, Kovac S, Hallmeyer-Elgner S, Winkler G, Springub J, Niedhammer M, Roth E, Eisensehr I, Berrouschot J, Arnold S, Schroder M, Beige A, Oertel WH, Strzelczyk A, Haag A, Reif PS, Hamer HM; LaLiMo Study Group. The LaLiMo Trial: lamotrigine compared with levetiracetam in the initial 26 weeks of monotherapy for focal and generalised epilepsy--an open-label, prospective, randomised controlled multicenter study. J Neurol Neurosurg Psychiatry. 2012 Nov;83(11):1093-8. doi: 10.1136/jnnp-2011-301999. Epub 2012 May 17. PMID 22595362